CLINICAL TRIAL: NCT02063555
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Multiple-Dose, Dose-Ranging Study of the Safety and Immunogenicity of DAR-901, a Killed, Non-Tuberculous Mycobacterial Vaccine, in HIV-negative and HIV-positive Adults Who Have Previously Received BCG
Brief Title: Phase I Trial of DAR-901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAR-901-MDES
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; BCG; HIV; TB Vaccines
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DAR-901 (Experimental): Intradermal administration at 0, 2 and 4 months
  Three dose groups in dose escalation: 0.1 mg, 0.3 mg and 1.0 mg, all constituted in 0.1 mL
  Interventions: Biological: DAR-901
- BCG (Active Comparator): Intradermal injection of 0.1 mL saline at 0 mos, 2 mos, intradermal injection of 0.1 mL BCG at 4 mos
  Interventions: Biological: BCG
- Sterile saline (Placebo Comparator): Intradermal injection of 0.1 mL sterile saline at 0, 2 and 4 mos
  Interventions: Biological: Sterile saline

INTERVENTIONS:
Biological: DAR-901
  Arms: DAR-901
Biological: BCG
  Arms: BCG
Biological: Sterile saline
  Arms: Sterile saline

SUMMARY:
This is a Phase 1, randomized, controlled, double-blind, multiple-dose, dose-ranging study of DAR 901, (an inactivated whole cell mycobacterial vaccine) to be conducted in HIV negative and HIV positive adults previously vaccinated with BCG. The goals of the trial are to determine the safety, tolerability, and immunogenicity of multiple doses of the vaccine at different dose levels, ranging from 0.1 to 1 mg.

ELIGIBILITY:
Inclusion Criteria:

All subjects: age 18-65, prior BCG vaccine (scar)

56 HIV negative subjects: negative ELISA for HIV (48 subjects with negative IGRA, 8 subjects with positive IGRA)

21 HIV positive subjects: positive ELISA for HIV, on ART (13 subjects with negative IGRA, 8 subjects with positive IGRA)

Exclusion Criteria: pregnancy, positive serology for hepatitis B or C, active tuberculosis immunosuppression, severe medical illness

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety | 10 months
  Subjects will be followed for both systemic side effects and injection site reactions

SECONDARY OUTCOMES:
Immunogenicity | 10 months
  Cellular and humoral responses to the vaccine antigen will be tested at baseline and after each of 3 doses of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. von Reyn, MD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Masonou T, Hokey DA, Lahey T, Halliday A, Berrocal-Almanza LC, Wieland-Alter WF, Arbeit RD, Lalvani A, von Reyn CF. CD4+ T cell cytokine responses to the DAR-901 booster vaccine in BCG-primed adults: A randomized, placebo-controlled trial. PLoS One. 2019 May 23;14(5):e0217091. doi: 10.1371/journal.pone.0217091. eCollection 2019. PMID 31120957
- [Derived] Craig SR, Lahey T, Dixit A, Fordham von Reyn C. Altruism, Scepticism, and collective decision-making in foreign-born U.S. residents in a tuberculosis vaccine trial. BMC Public Health. 2018 Apr 23;18(1):535. doi: 10.1186/s12889-018-5460-3. PMID 29685114
- [Derived] von Reyn CF, Lahey T, Arbeit RD, Landry B, Kailani L, Adams LV, Haynes BC, Mackenzie T, Wieland-Alter W, Connor RI, Tvaroha S, Hokey DA, Ginsberg AM, Waddell R. Safety and immunogenicity of an inactivated whole cell tuberculosis vaccine booster in adults primed with BCG: A randomized, controlled trial of DAR-901. PLoS One. 2017 May 12;12(5):e0175215. doi: 10.1371/journal.pone.0175215. eCollection 2017. PMID 28498853